CLINICAL TRIAL: NCT07368803
Title: Evaluation of the Safety, Tolerability and Efficacy of iNeo-Vac-R01, an Individualized mRNA Therapeutic Technology Based on Tumor Neoantigens, for Adjuvant Treatment in Patients With Biliary Malignant Tumors After Radical Resection
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yifan Wang (Other)
Collaborators: Hangzhou Neoantigen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yifan Wang, Chief Physician，Director，Principal Investigator, Sir Run Run Shaw Hospital
Organization: Sir Run Run Shaw Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-2714-01
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Biliary Malignant Tumors

STUDY DESIGN:
Intervention Model Description: Interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group (Experimental): Personalized mRNA Vaccine iNeo-Vac-R01
  Interventions: Biological: iNeo-Vac-R01

INTERVENTIONS:
Biological: iNeo-Vac-R01 — IH injection

SUMMARY:
The primary objective of this study is to evaluate the safety of iNeo-Vac-R01, an individualized mRNA therapeutic technology based on tumor neoantigens, for the adjuvant treatment of patients with biliary malignant tumors after radical resection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, >/= 18 years old and </= 75 years old；
2. Biliary malignant tumors confirmed by histopathological or cytological examination that are eligible for radical resection；
3. Subjects must have one of the histologically- or cytologically-confirmed advanced (locally advanced or metastatic) digestive system neoplasms, have measurable disease at study entry defined by RECIST v1.1. Subjects must have tumor progression after standard treatment or are intolerant or are unwilling to receive standard treatment. The toxic effects of previous anti-tumor treatments have returned to </= grade 1 defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 or to the level specified by the inclusion/exclusion criteria.
4. Expected survival >/= 6 months.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 ~ 1；
6. Sufficient tumor tissue samples can be obtained from subjects for genetic analysis, with at least 2 puncture tissues with a tumor purity of ≥ 50% required for puncture samples and at least 0.5cm of tissue required for surgical samples. Alternatively, the original gene sequencing data required for tumor neoantigen analysis can be provided, including full exon sequencing data of tumor tissue, transcriptome sequencing data, and full exon sequencing data of peripheral blood；
7. Echocardiographic evaluation: left ventricular ejection fraction (LVEF) >/= 50%.
8. The organ function level must meet the following requirements: absolute neutrophil count (ANC) >/= 1.5 × 10^9/L, platelet count (PLT) >/= 80 × 10^9/L, hemoglobin (Hb) >/= 90 g/L; serum total bilirubin (TBIL) </= 1.5 × ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) </= 2.5 × ULN (if there is liver metastasis, TBIL </= 3 × ULN, AST, ALT </= 5 ×ULN are allowed), serum albumin >/= 28g/L, serum creatinine </= 1.5 × BUN, Glomerular filtration rate >/= 50mL/min, prothrombin time (PT) and activated partial thromboplastin time (APTT) and international standardized ratio (INR) </= 1.5 × ULN (without anticoagulant therapy) .
9. For women of childbearing potential: having a negative serum or urine pregnancy test within 7 days prior to study initiation, agreement to remain abstinent or use contraceptive measures during the treatment period.
10. For men: agreement to remain abstinent or use contraceptive measures during the treatment period.
11. Able to comply with the study protocol and follow-up procedures.
12. Voluntarily participate in the study and sign the informed consent form. If a subject is unable to read the informed consent form (e.g., illiterate subjects), a witness shall be present to observe the informed consent process and sign the informed consent form on their behalf.

Exclusion Criteria:

1. Subjects with cancer requiring anti-tumor treatment within the 5 years prior to enrollment in the study (except stage I prostate cancer, cervical cancer in situ, breast cancer in situ, papillary thyroid cancer and non-melanoma skin cancer that have been treated).
2. Subjects who received major surgery, or had obvious traumatic injury or long-term untreated wounds or fractures within 2 weeks prior to the first dose of iNeo-Vac-R01.
3. Subjects whose sequencing data was found that there are no new antigens available for individualized immunotherapy after analysis.
4. Subjects who prepare to undergo or have previously received bone marrow transplantation, allogeneic organ transplantation, or allogeneic hematopoietic stem cell transplantation. Subjects who receive other anti-tumor treatments within 2 weeks prior to the first dose of iNeo-Vac-R01, including surgical treatment, chemotherapy, radiation therapy, targeted therapy, endocrine therapy, immunotherapy, biological therapy, interventional therapy, or other clinical trial related treatments.
5. Subjects who need to use immunosuppressants, or systemic or absorbable local glucocorticoids therapy to achieve immunosuppressive effects and continue to use them within 7 days before the first administration (excluding those with daily doses of glucocorticoids less than 10mg of prednisone or doses of other therapeutic glucocorticoids equal to 10mg of prednisone).
6. Subjects with symptomatic or untreated central nervous system metastases, except those underwent complete resection and/or radiotherapy and proven to be stable or improved (confirmed to be stable or improved for at least 4 weeks before the first dose of iNeo-Vac-R01 by CT or MRI, with no evidence of brain edema and no need for glucocorticoids or anticonvulsants.
7. Subjects who received other vaccines within 4 weeks before the first dose of iNeo-Vac-R01, and are expected to receive other vaccines during treatment period of the study or within 60 days after the last dose of iNeo-Vac-R01.
8. Subjects who have an active infection or uncontrollable infection requiring systemic treatment, including fungi, bacteria, viruses, or other infections; subjects with active tuberculosis;
9. Subjects with positive hepatitis B surface antigen (HBsAg) and/or positive hepatitis B core antibody (HBcAb) and positive hepatitis B virus DNA titer detection greater than normal range; positive hepatitis C virus (HCV) antibody and HCV RNA detection greater than normal range; positive human immunodeficiency virus antibody; positive treponema pallidum-specific antibody.
10. Subjects with autoimmune diseases or immune deficiencies treated with immunosuppressive drugs, except vitiligo, type 1 diabetes, autoimmune hypothyroidism requiring hormone treatment and psoriasis not requiring systemic treatment; known history of primary immunodeficiency.
11. Subjects with cardiocerebrovascular events: previously or currently heart valve disease >/= grade 3, heart failure within 8 weeks before the first dose of iNeo-Vac-R01 (New York Heart Association [NYHA] cardiac function >/= grade II, myocardial infarction, unstable angina, stroke, transient ischemic attack, cardiac surgery (including coronary artery bypass grafting or percutaneous coronary intervention) within 8 weeks before the first dose of iNeo-Vac-R01, concomitant severe electrocardiogram abnormalities (such as ventricular flutter, ventricular fibrillation, multiform ventricular tachycardia, sick sinus syndrome, third degree atrioventricular block without pacemaker treatment, QTc >/= 480ms, and other conditions evaluated by the investigators as severe abnormalities), hypertension with poor drug control (systolic blood pressure >/= 160mmHg and/or diastolic blood pressure >/= 100mmHg), or other cardiocerebrovascular diseases that have been evaluated by the investigators as unsuitable for participation in this trial.
12. Subjects with respiratory disease: previously or currently pulmonary fibrosis, interstitial lung disease, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe asthma, pulmonary hypertension or severe impairment of lung function, etc.
13. Subjects with moderate to severe ascites with clinical symptoms; uncontrolled or moderate to equal amounts of pleural effusion and pericardial effusion.
14. Subjects with drug abuse; clinical or psychological or social factors that affect informed consent or research implementation.
15. Subjects with a history of allergies to immunotherapy or vaccines, or other potential immunotherapy allergies identified by the investigators.
16. Subjects identified that it is not suitable for enrollment or may not be able to complete this experiment for other reasons by the investigators.
17. Vulnerable groups, including individuals with mental illness, cognitive impairment, critical patients, minors, pregnant or lactating women, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose for Safety and Tolerability Evaluation | 21 days after last iNeo-Vac-R01 dose
  Based on the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, the number of subjects with adverse events and/or dose-limiting toxicities will be counted as indicators for evaluating the safety and tolerability dose of iNeo-Vac-R01 Injection. The safety data collection visit will be conducted at 21 days after the last treatment administration.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years after first dose of iNeo-Vac-R01
  OS is defined as time between the date of the first dose of iNeo-Vac-R01 and the date of death due to any cause.
Relapse-Free Survival (RFS) | 3 years after first dose of iNeo-Vac-R01
  The time from the date of the first administration of iNeo-Vac-R01 Injection to the date of disease recurrence or death from any cause. The assessment duration is 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Institute of Minimally Invasive Surgery, Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No